CLINICAL TRIAL: NCT07021365
Title: Comparison of Ganglion Impar Radiofrequency Ablation and Phenol Neurolysis Techniques for Chronic Coccydynia Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.2024.1470
Record Dates: First submitted 2025-05-29; First posted 2025-06-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Coccygodynia; Coccydynia
Keywords: coccygodinia; chronic; radiofrequency ablation; phenol neurolysis; coccydynia
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Phenol; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ganglion Impar Radiofrequency Ablation (Active Comparator)
  Interventions: Device: Radiofrequency ablation alone
- Ganglion Impar Phenol Neurolysis (Active Comparator)
  Interventions: Drug: Phenol Injection

INTERVENTIONS:
Drug: Phenol Injection — n patients diagnosed with chronic coccydynia, a ganglion impar block is initially performed following conservative treatment. In cases where this intervention provides limited benefit, ganglion impar phenol neurolysis is performed. A short-acting local anesthetic (3-4 mL of 1% prilocaine) will be administered into the skin and subcutaneous tissues. A 90 mm 22-gauge Quincke-tipped spinal needle will be advanced via the trans-coccygeal route under fluoroscopic guidance with intermittent imaging. The needle's position in the area anterior to the coccyx, where the ganglion impar is located, will be confirmed using 1-2 mL of contrast agent (iohexol). If the desired spread of contrast is observed, 5 mL of 7% phenol will be injected.
  Arms: Ganglion Impar Phenol Neurolysis
Device: Radiofrequency ablation alone — In patients diagnosed with chronic coccydynia, a ganglion impar block is initially performed following conservative treatment. In cases where this intervention provides limited benefit, ganglion impar radiofrequency (RF) ablation-routinely used in clinical practice-will be performed by an experienced pain specialist (SŞ) with at least 10 years of expertise in this procedure.
  Using fluoroscopic guidance and intermittent imaging, a 100 mm RF cannula with an injection tube will be advanced trans-coccygeally. After confirming the needle's position at the site of the ganglion impar in front of the coccyx with 1-2 mL of contrast agent (iohexol), sensory stimulation will be applied via the RF generator to confirm that the needle tip is at the patient's pain site. Motor stimulation will also be performed to ensure there is no muscle contraction. At this stage, 2 mL of lidocaine will be administered before initiating ablation at 80°C for 90 seconds.
  Arms: Ganglion Impar Radiofrequency Ablation

SUMMARY:
Radiofrequency ablation and phenol neurolysis of the ganglion impar are methods used in cases unresponsive to medication, particularly in patients who derive short-term or partial relief from the initial ganglion impar block. In clinical practice, clinicians frequently use these two injections in patients with treatment-resistant pain who only partially benefit from the initial blockade procedure.

To date, the medical literature lacks a comprehensive study comparing the efficacy of radiofrequency ablation and phenol neurolysis in patients who partially benefit from ganglion impar block. Therefore, this study is designed to compare the effectiveness of these two methods in patients with chronic coccydynia.

DETAILED DESCRIPTION:
Ganglion impar radiofrequency ablation and phenol neurolysis are treatment options for patients who do not respond to medication, especially those experiencing only temporary or partial relief from an initial ganglion impar block. In clinical practice, these two injection techniques are commonly employed in managing persistent pain in such cases.

Radiofrequency Ablation (RFA):

This technique aims to eliminate pain by thermally damaging the nerves that carry pain sensations. Under real-time imaging guidance, a radiofrequency needle is advanced through the intervertebral disc from the tailbone region to the anatomical area called the ganglion impar. The needle tip location is confirmed with contrast dye. At this point, motor and sensory stimulation is applied to ensure the needle is not affecting motor function and to identify the site where the pain stimulus matches the patient's complaint. Once confirmed, heat application is initiated. Prior to heat delivery, a local anesthetic is administered to ensure the procedure is painless.

Phenol Neurolysis:

This method aims to chemically destroy the nerves carrying pain signals from the coccyx area using phenol. The procedure is performed similarly to RFA: a radiofrequency needle is inserted through the disc between spinal bones under real-time imaging guidance to reach the ganglion impar. After confirming the needle position with contrast dye, a local anesthetic is administered, and then phenol is applied to chemically ablate the sensory fibers without pain.

No major complications have been reported in the literature regarding these two procedures. However, minor complications may occur, such as vasovagal reactions (temporary fainting), minor bleeding, infection, and vascular injection.

Study Design:

The study will include patients under the care of the Marmara University Pain Medicine Department who have not responded to medication and have received short-term or partial benefit from an initial ganglion impar block. These patients will be randomly assigned via computer software into two groups. One group will undergo the radiofrequency ablation procedure described above, and the other group will receive phenol neurolysis. The patients will be followed for six months, and the effectiveness of these two widely used but yet-to-be-compared treatments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Presence of chronic coccydynia lasting at least 3 months
* Pre-procedural pain score of 4 or higher on the Numeric Rating Scale (NRS)
* Patients who have undergone a ganglion impar block within the last 3 months and experienced limited benefit (i.e., less than 50% reduction in pain compared to pre-treatment) and/or short-term relief (less than 4 weeks)

Exclusion Criteria:

* History of surgery involving the sacrococcygeal region
* Prior treatment with ganglion impar phenol neurolysis or radiofrequency ablation
* Coagulopathies (bleeding disorders)
* Infection
* Spondylolisthesis, scoliosis, or lumbar spinal stenosis
* Malignancy
* Pregnancy
* History of allergic reaction to the administered injectates
* History of major psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale-11 | Treatment to 6 months post-treatment
  A subjective outcome measure to assess pain (Min:0 Max:10). Higher scores indicate more severe pain.

SECONDARY OUTCOMES:
Short Form-12 Health Survey | Treatment to 6 months post-treatment.
  The SF-12 (Short Form-12 Health Survey) is a validated instrument used to evaluate health-related quality of life, with scores ranging from 0 to 100. Higher scores reflect better overall health status.
Douleur Neuropathique 4 | Treatment to 6 months post-treatment.
  The DN4 (Douleur Neuropathique 4) questionnaire is a diagnostic screening tool designed to detect the presence of neuropathic pain, with scores ranging from 1 to 10. Higher scores suggest a greater probability of neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Sagir O, Demir HF, Ugun F, Atik B. Retrospective evaluation of pain in patients with coccydynia who underwent impar ganglion block. BMC Anesthesiol. 2020 May 11;20(1):110. doi: 10.1186/s12871-020-01034-6. PMID 32393277
- [Background] Demircay E, Kabatas S, Cansever T, Yilmaz C, Tuncay C, Altinors N. Radiofrequency thermocoagulation of ganglion impar in the management of coccydynia: preliminary results. Turk Neurosurg. 2010 Jul;20(3):328-33. doi: 10.5137/1019-5149.JTN.2852-09.0. PMID 20669105
- [Background] Howard PD, Dolan AN, Falco AN, Holland BM, Wilkinson CF, Zink AM. A comparison of conservative interventions and their effectiveness for coccydynia: a systematic review. J Man Manip Ther. 2013 Nov;21(4):213-9. doi: 10.1179/2042618613Y.0000000040. PMID 24421634
- [Background] Kircelli A, Demircay E, Ozel O, Coven I, Isik S, Civelek E, Kabatas S. Radiofrequency Thermocoagulation of the Ganglion Impar for Coccydynia Management: Long-Term Effects. Pain Pract. 2019 Jan;19(1):9-15. doi: 10.1111/papr.12698. Epub 2018 May 16. PMID 29617062
- [Background] Sencan S, Kenis-Coskun O, Demir FGU, Cuce I, Ercalik T, Gunduz OH. Ganglion Impar block improves neuropathic pain in coccygodynia: A preliminary report. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):612-617. doi: 10.1016/j.pjnns.2018.08.006. Epub 2018 Aug 28. PMID 30195465
- [Background] Karadimas EJ, Trypsiannis G, Giannoudis PV. Surgical treatment of coccygodynia: an analytic review of the literature. Eur Spine J. 2011 May;20(5):698-705. doi: 10.1007/s00586-010-1617-1. Epub 2010 Nov 3. PMID 21046173